CLINICAL TRIAL: NCT05255380
Title: Pilot Randomized Controlled Trial Examining the Effects of Daily Mindfulness in Woman With a History of Child Adversity
Brief Title: Examine the Effects of Mindfulness in Woman With a History of Child Adversity
Acronym: EMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB# 21-35255; R00AG062778 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-02-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Stress; Psychological Stress; Child Maltreatment; Depressive Symptoms; Signs and Symptoms
Keywords: Mindfulness; Adverse childhood experiences; Stress; Depressive symptoms
MeSH Terms: conditions — Stress, Psychological; Depression; Signs and Symptoms | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either a Mindful Activity group or a Mindful Awareness group. Randomization will occur by chance (50%) at the end of the baseline visit.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Activity group (Experimental): Participants complete mindfulness and compassion-based practices via the study app.
  Interventions: Behavioral: Mindfulness and compassion-based practices; approximately 5-10 minutes two times/day
- Mindful Awareness group (Sham Comparator): Participants monitor and report their thoughts and feelings via the study app.
  Interventions: Behavioral: Mindful awareness and reporting of current thoughts and feelings, 2 times/day

INTERVENTIONS:
Behavioral: Mindfulness and compassion-based practices; approximately 5-10 minutes two times/day — The app-based (audio-guided) interventions consist of mindfulness and compassion-based practices that are selected to maximize their effect on stress targets. Interventions include, for example, practices that focus on the breath/body (e.g., 3-minute breathing space; compassionate body scan; five senses mediation), on increasing participants' inner resources (e.g., imaging a safe person or safe place), on reducing negative affect (e.g., self-compassion and acceptance-based practices), or on increasing positive emotions (e.g., gratitude practice; metta practices).
  Arms: Mindful Activity group
Behavioral: Mindful awareness and reporting of current thoughts and feelings, 2 times/day — Participants are instructed to be mindful (pay attention) to their current thoughts and feelings and complete ecological momentary assessments of their current psychological stress states (e.g., stress appraisals, affect, perseverative cognitions, self-criticism, social connection)
  Arms: Mindful Awareness group

SUMMARY:
The aim of this pilot Randomized Controlled Trial (RCT) is to test whether brief mindfulness-based practices will improve well-being and health in women (age 30-50) with a history of early life adversity. Following a baseline visit (remotely via Zoom), participants are randomized (50% probability) to either a Mindful Activity group or a Mindful Awareness group. In the Mindful Activity group, participants will complete brief (approximately 5-10 min) audio-guided mindfulness practices twice a day (morning and evening) for 8 weeks using the study app. This is followed by a brief survey about their current thoughts and feelings. In the Mindful Awareness group, participants are asked to be mindful (pay attention) to their thoughts and feelings twice a day (morning and evening) for 8 weeks using the study app. After the 8-week intervention period, all participants complete a follow-up visit (remotely). Primary goals of the pilot RCT are to test acceptability, feasibility, and adherence.

DETAILED DESCRIPTION:
The pilot Randomized Controlled Trial (RCT) randomly assigns midlife women (age 30-50) with a history of early life adversity to either a Mindful Activity group or a Mindful Awareness group to primarily test acceptability, feasibility, and adherence. Randomization will occur by chance at the end of the baseline visit.

Participants randomized to the Mindful Activity group will receive 8 weeks of ecological momentary assessment and intervention sessions via the study app. Mindfulness-based interventions consist of mindfulness and compassion-based practices. For example, practices focus on the breath/body (e.g., 3-minute breathing space; compassionate body scan; five senses mediation), on increasing participants' inner resources (e.g., imaging a safe person or safe place), on reducing negative affect (e.g., self-compassionate and acceptance-based practices), or on increasing positive emotions (e.g., gratitude practice; metta practices). All interventions are audio-guided and approximately 5-10 minutes. Participants complete two mindfulness interventions/day (one in the morning; one in the evening). After completing a mindfulness-based intervention, participants will complete ecological momentary assessments of their current psychological stress states (e.g., stress appraisals, affect, perseverative cognitions, self-criticism, social connection) via the study app.

Participants randomized to the Mindful Awareness group are instructed to be mindful (pay attention) to their current thoughts and feelings and complete ecological momentary assessments of their current psychological stress states (e.g., stress appraisals, affect, perseverative cognitions, self-criticism, social connection) twice/day (morning and evening) for 8 weeks via the study app.

A trained research assistant will monitor participant adherence and address potential difficulties. All participants will complete assessments at baseline (pre-intervention) and post-intervention (after the 8-week intervention). Weekly measures of depressive symptoms are also obtained. The investigators plan to consent about 100 participants with the goal of having 70 eligible participants enrolled in the study (about 35 in each group).

ELIGIBILITY:
Inclusion Criteria:

1. female sex and gender identity (to control for sex and gender differences in stress responses and health outcomes)
2. age 30-50 (to examine intervention effects on health outcomes in midlife)
3. ≥2 Adverse Childhood Experiences (to ensure exposure to early life adversity)
4. mild depressive symptoms (to allow for outcome improvements: PHQ-9 ≥ 5)
5. having a smartphone (to access app-based assessments/interventions)

Exclusion Criteria:

1. Non-English speaker or unable to provide informed consent
2. Current regular mindfulness practice (exclude if >20 min/week)
3. Major psychiatric condition, including psychosis/schizophrenia, bipolar disorder, post-traumatic stress disorder, eating disorders, alcohol/substance use, major depression (PHQ-9 ≥ 15), and self-harm or suicidal ideation
4. Major medical conditions, including no history of coronary heart disease, diabetes, severe asthma or lung disease, autoimmune disorders, infectious disease, epilepsy, brain injury, endocrine disorders, diagnosis of cancer or chemotherapy or radiation in the past 10 years
5. Free from medications known to affect the immune and endocrine systems with the exception of antidepressant medication and oral contraceptives
6. Psychotherapy treatment permitted if stable (≥3 months)
7. Current smoking and nicotine use
8. Currently pregnant

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity.
Enrollment: 72 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention will be measured with an adapted version of the Treatment Acceptability Questionnaire (TAQ). | Assessed at post-intervention, approximately 8 weeks from baseline
  The Treatment Acceptability Questionnaire (TAQ) is a six-item scale assessing whether participants view their assigned intervention as acceptable, ethical, and effective. Items are rated on a 7-point Likert scale (e.g., 1 "very unacceptable" to 7 "very acceptable), with a possible score range from 6 to 42. Higher scores indicate better treatment acceptability and positive perceptions of the treatment. A total mean score of at least 24 will indicate sufficient acceptability of the intervention.
Feasibility, as indicated by numbers of participants screened (completed web-based screener and phone screener), eligible based on web-based screener and phone screener, consented, randomized to treatment, and retained at follow-up. | Anticipated study period of 12 months
  Feasibility outcomes will include: >70% of eligible participants (passed web-based and phone screener) will be consented, >70% of consented participants will pass further baseline screening procedures and will be randomized to treatment, >70% of participants who are randomized to treatment will be retained at follow-up. Reasons for ineligibility and drop out will also be assessed.
Adherence, as measured by the percentage of assigned and completed intervention group practices. | Baseline to follow-up, an anticipated 8 weeks
  Completion of at least 50% of assigned intervention group practices (Ecological Momentary Assessments for Mindful Awareness group; mindfulness practices for Mindful Activity group) is considered acceptable.

SECONDARY OUTCOMES:
Change in depressive symptoms, as measured by the total score on the 9-item Patient Health Questionnaire (PHQ-9). | Baseline to post-intervention, an anticipated 8 weeks
  The 9-item Patient Health Questionnaire (PHQ-9) has a total score scale range of 0 to 27, with higher values indicating more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie E Mayer, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No